CLINICAL TRIAL: NCT02362958
Title: Sun Yat-sen University Cancer Center
Brief Title: A Multi-Center Study of Lapatinib in Patients With Trastuzumab-refractory Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhong-yu Yuan, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-005
Record Dates: First submitted 2015-02-08; First posted 2015-02-13 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: HER2 Positive Breast Cancer
MeSH Terms: interventions — Lapatinib; Capecitabine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lapatinib and Capecitabine or Vinorelbine (Experimental): Lapatinib 1250mg qd and Capecitabine 1000mg/m2 bid or Vinorelbine 25mg/m2 iv (d1,d8)
  Interventions: Drug: lapatinib and capecitabine or vinorelbine

INTERVENTIONS:
Drug: lapatinib and capecitabine or vinorelbine — lapatinib 1250 mg qd and Capecitabine 1000 mg/m2 bid or Vinorelbine 25mg/m2(d1,d8)
  Other Names: Tykerb; Xeloda;NVB

SUMMARY:
Evaluating the Efficacy of Lapatinib in Combination With Chemotherapy in Patients With Trastuzumab-refractory Metastatic HER2-positive Breast Cancer.

DETAILED DESCRIPTION:
Some studies has demonstrated that even in trastuzumab pretreated patients with HER-2 positive breast cancer, might benefit from the treatment of trastuzumab. However, there is small benefit for some patients having short disease-free survival after adjuvant trastuzumab or short progression-free survival after first-line trastuzumab-based therapy. In clinical practice, the investigators also found it is fact. And the investigators have a scientific rationale for clinical testing of lapatinib plus chemotherapy in patients with trastuzumab-refractory, metastatic HER2-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic breast cancer
* Eastern Cooperative Oncology Group (ECOG) 0 or 1
* HER2-expressing primary or metastatic tumor
* Recurrence within 1 year completing adjuvant trastuzumab OR rapid progress following first-line trastuzumab-based care.
* Measurable disease with Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Normal organ function, including bone marrow function, renal function, liver function, and cardiac function
* Signed and dated an informed consent form
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* Pregnant or breast feeding
* left ventricular ejection fraction (LVEF) < 45% by echocardiogram
* Disease-free interval (DFI) less than 12 months
* Uncontrolled medical problems
* Any previous malignancy exceptions for carcinoma of the cervix, squamous carcinoma of the skin, or basal cell carcinoma of the skin
* Patients were unable or unwilling to comply with program requirements

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2015-01-09 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 36 months
  The time from randomization to disease progression or death from any causes

CONTACTS AND LOCATIONS:
Overall Officials: Zhong-Yu Yuan, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duan F, Zhong M, Ma Y, Song C, Zhang L, Lin Y, Wu Z, Zhang Y, Huang J, Xu F, Shi Y, Wang S, Yuan Z, Xia W, Bi X. The efficacy of human epidermal growth factor receptor 2 (HER2) blockade switching mode in refractory patients with HER2-positive metastatic breast cancer: a phase II, multicenter, single-arm study (SYSUCC-005). BMC Cancer. 2022 Mar 15;22(1):271. doi: 10.1186/s12885-022-09399-2. PMID 35291977